CLINICAL TRIAL: NCT03518242
Title: Defining the Molecular Profile of Breast Cancer in Uganda and Its Clinical Implications
Brief Title: Molecular Profile of Breast Cancer in Ugandan Patients With Stage IIB-III Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U025; NCI-2018-02609 (Registry Identifier: NCI / CTRP); RG1001403 (Other: Fred Hutch/University of Washington Cancer Consortium); 8424 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2018-04-25; First posted 2018-05-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Breast Cancer Female; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Invasive Breast Carcinoma; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8
MeSH Terms: interventions — Cyclophosphamide; Methotrexate; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (Specimen collection, chemotherapy) (Experimental): SPECIMEN COLLECTION: Patients undergo collection of tumor tissue and peripheral blood samples for analysis via next generation sequencing to identify novel pathways in the pathogenesis of breast cancer.
  TREATMENT: Patients are invited to participate in a treatment study. Patients receive cyclophosphamide PO daily on days 1-21, methotrexate PO QD on days 1, 8, and 15, and capecitabine PO BID on days 1-14. Treatment repeats every 21 days for 8 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Methotrexate; Drug: Capecitabine; Procedure: Biospecimen Collection

INTERVENTIONS:
Drug: Cyclophosphamide — Given PO
  Other Names: Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclostin; Fosfaseron; Mitoxan; Neosar
Drug: Methotrexate — Given PO
  Other Names: Abitrexate; Brimexate; Emtexate; Fauldexato; Ledertrexate; Medsatrexate; Methylaminopterin
Drug: Capecitabine — Given PO
  Other Names: Xeloda
Procedure: Biospecimen Collection — Undergo biospecimen collection

SUMMARY:
This phase I trial studies the molecular profile of breast cancer in Ugandan patients with stage IIB-III breast cancer. Creating a molecular profile of breast cancer my help doctors learn more about biological factors associated with breast cancer in Ugandan patients with as well as measure the benefits of locally available diagnostic studies and the possibility of providing treatment via oral medication.

DETAILED DESCRIPTION:
OUTLINE:

SPECIMEN COLLECTION: Patients undergo collection of tumor tissue and peripheral blood samples for analysis via next generation sequencing to identify novel pathways in the pathogenesis of breast cancer.

TREATMENT: Patients are invited to participate in a treatment study. Patients receive cyclophosphamide orally (PO) daily on days 1-21, methotrexate PO QD on days 1, 8, and 15, and capecitabine PO twice daily (BID) on days 1-14. Treatment repeats every 21 days for 8 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study, patients are followed up for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Women with any menopausal status, with newly diagnosed, locally advanced and histologically confirmed invasive breast cancer (Patients with stage 2B [i.e. T3N0], 3A, 3B, and 3C disease)
* Absolute neutrophil count (ANC) > 1500/mm
* Hemoglobin > 9 g/dL
* Platelets >=100,000 cells/mm^3
* Total bilirubin =< 1.2 mg/dL
* International normalized ratio (INR) =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 1.5 x ULN
* Serum alkaline phosphatase should be 1.5 x ULN
* Patients with positive hepatitis B or C serologies without known active disease must meet the eligibility requirements for ALT, AST, total bilirubin, INR, activated partial thromboplastin time (aPTT), and alkaline phosphatase on at least two consecutive occasions, separated by at least 1 week
* Adequate renal function with serum creatinine < 1.5 x ULN
* Premenopausal patients must have a negative serum or urine pregnancy test, including women who have had a tubal ligation and for women less than 12 months after the onset of menopause
* Women of childbearing potential must be willing to use one highly effective form of nonhormonal contraception or two effective forms of nonhormonal contraception by the patient and/or partner and continue its use for the duration of the study treatment
* Left ventricular ejection fraction >= 50%
* Eastern Cooperative Oncology Group (ECOG) performance status < 2
* Signed written informed consent

Exclusion Criteria:

* A treatment-free interval of < 6 months with previous chemotherapy
* Active, unresolved infection or systemic disease (e.g. pulmonary or metabolic disease)
* Patients with active liver disease
* Patients with active cardiac disease, including congestive heart failure (or therapy specifically for congestive heart failure [CHF])
* Patients with uncontrolled hypertension (diastolic >100 mmHg or systolic > 160 mmHg)
* Known hypersensitivity to any of the drugs
* Significant current illness (including psychiatric illness)
* Any social situations or other conditions that in the opinion of the investigator limit compliance with study requirements
* Calcium imbalance
* Patients that have received treatment with sorividine or brividine (herpex) or any related analogue within 4 weeks prior to starting the investigational product (IP)
* Eye problems
* Patients on any of the following medications: acitretin, azathioprine, Bacillus Calmette Guerin (BCG) (intravesicular), belimumab, deferiprone, diphyrone, etanercept, foscarnet, gimeracil, levetriracetam, natalizumab, pimercrolimus, retinoids, sulfazalazine, tacrolimus tofacitininb
* Patients receiving any anticoagulation (including warfarin)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-04 (Actual)

PRIMARY OUTCOMES:
Distribution of molecular subtypes | Up to 9 months
  Will classify Ugandan women into four categories based on molecular subtypes: estrogen receptor (ER) negative (-)/progesterone receptor (PR) - /HER2 - (triple negative), ER-/PR-/HER positive (+) (HER2), ER+/PR+/HER2- (luminal A), and ER/PR+/HER2 + (luminal B) and compare to aggregate data from previously published data on a cohort of African-American women using chi square tests.
Sensitivity to polymerase chain reaction (PCR) | Up to 9 months
  Sensitivity, defined as the proportion of women with a particular receptor detected by PCR, among those women who had the receptor detected by immunohistochemistry (IHC), to polymerase chain reaction (PCR) will be estimated with 95% confidence intervals (CIs), using IHC as the gold standard. Will also calculate the percent agreement between PCR and IHC, and compute the kappa statistic with 95% CIs to assess receptor status agreement between reverse transcription (RT)-PCR and IHC.
Specificity of PCR | Up to 9 months
  Specificity, defined as the proportion of women with a receptor not detected by PCR, among women who did not have the receptor detected by IHC, to PCR will be estimated with 95% CIs, using IHC as the gold standard. Will also calculate the percent agreement between PCR and IHC, and compute the kappa statistic with 95% CIs to assess receptor status agreement between RT-PCR and IHC.
Patient adherence to treatment | Up to 168 days (8 cycles)
  Patient adherence as the proportion of women completing 8 cycles of therapy compared to historical controls from the UCI cancer registry database using chi square tests
Incidence of adverse events | Up to 6 months
  Will describe the extent of adverse events assessed using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0. Will also compare patient adherence and adverse events using chi square tests and compare survival using log-rank tests.
Overall Survival | Up to 1 year
  Will use Kaplan-Meier methodology.

CONTACTS AND LOCATIONS:
Overall Officials: Manoj Menon, Principal Investigator — Fred Hutchinson Cancer Center
Locations (2):
- Uganda (2):
  - New Mulago Hospital, Kampala
  - Uganda Cancer Institute, Kampala

IPD SHARING:
Plan to Share IPD: No